CLINICAL TRIAL: NCT04214392
Title: A Phase 1 Study to Evaluate Chimeric Antigen Receptor (CAR) T Cells With a Chlorotoxin Tumor-Targeting Domain for Patients With MMP2+ Recurrent or Progressive Glioblastoma
Brief Title: Chimeric Antigen Receptor (CAR) T Cells With a Chlorotoxin Tumor-Targeting Domain for the Treatment of MMP2+ Recurrent or Progressive Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19309; NCI-2019-08393 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19309 (Other: City of Hope Medical Center)
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Glioblastoma; Recurrent Malignant Glioma; Recurrent WHO Grade II Glioma; Recurrent WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Chlorotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (CAR T cell therapy) I (Experimental): Arm 1 participants will undergo resection/biopsy of their tumor and placement of a Rickham catheter at the site of the resection/biopsy. Patients receive chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes NCI SYs via single delivery starting on day 0 for 3 weekly cycles over 28 days. Each treatment cycle begins with one CAR T cell infusion delivered intracranial intratumoral or intracavitary [ICT] and lasts for 1 week. Beginning 1 week after cycle 3, patients may continue with CAR T cell treatment per principal investigator and patient discretion. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes (via ICT delivery)
- Treatment (CAR T cell therapy) II (Experimental): Arm 2 participants will undergo resection/biopsy of their tumor and placement of a Rickham catheter at the site of the resection/biopsy and the lateral ventricle. Patients receive chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes NCI SYs via dual delivery starting on day 0 for 3 weekly cycles over 28 days. Each treatment cycle begins with two CAR T cell infusions (intracranial intratumoral or intracavitary [ICT]) and also into the lateral ventricle (intracranial intraventricular [ICV]) and lasts for 1 week. Beginning 1 week after cycle 3, patients may continue with CAR T treatment per principal investigator and patient discretion. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes (via ICT/ICV dual delivery)

INTERVENTIONS:
Biological: Chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes (via ICT delivery) — Given via ICT delivery
  Other Names: Chlorotoxin-CD28-CD3z-CD19t-expressing CAR T-cells
  Arms: Treatment (CAR T cell therapy) I
Biological: Chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes (via ICT/ICV dual delivery) — Given via ICT/ICV dual delivery
  Other Names: Chlorotoxin-CD28-CD3z-CD19t-expressing CAR T-cells
  Arms: Treatment (CAR T cell therapy) II

SUMMARY:
This phase I trial studies the side effects and best dose of chimeric antigen receptor (CAR) T cells with a chlorotoxin tumor-targeting domain in treating patients with MPP2+ glioblastoma that has come back (recurrent) or that is growing, spreading, or getting worse (progressive). Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the feasibility and safety of dual delivery of chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes NCI SYs (chlorotoxin [CLTX]-CAR T cells) for participants with MMP2+ recurrent or progressive glioblastoma.

II. Determine the maximum tolerated dose schedule (MTD) and a recommended phase 2 dosing plan (RP2D) for dual delivery of CLTX-CAR T cells for participants with MMP2+ recurrent or progressive glioblastoma.

SECONDARY OBJECTIVES:

I. Describe persistence, expansion, and phenotype of endogenous and CLTX-CAR CAR T cells in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF).

II. Describe cytokine levels in PB, TCF, and CSF over the study period.

III. In research participants who receive the full schedule of 3 cycles of CLTX-CAR T cells:

IIIa. Estimate the six month progression free survival (PFS) rate. IIIb. Estimate the nine month overall survival (OS) rate. IIIc. Estimate disease response rates. IIId. Estimate median overall survival (OS).

IV. In study participants who undergo an additional biopsy/resection or autopsy:

IVa. Evaluate CAR T cell persistence in the tumor tissue and the location of the CAR T cells with respect to the injection site.

IVb. Evaluate CLTX-targeted antigen expression levels on tumor tissue pre and post CAR T cell therapy.

V. Use mathematical modeling of tumor growth to evaluate benefit of treatment.

OUTLINE: This is a dose-escalation study.

Patients receive chlorotoxin (EQ)-CD28-CD3zeta-CD19t-expressing CAR T-lymphocytes NCI SYs via dual delivery starting on day 0 for 3 weekly cycles over 28 days. Each treatment cycle begins with one or two CAR T cell infusions (one at each catheter site) and lasts for 1 week. Beginning 1 week after cycle 3, patients may continue with CAR T treatment per principal investigator and patient discretion. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 3, 6, 9, and 12 months, and then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative. Assent, when appropriate, will be obtained per institutional guidelines. Note: For research participants who do not speak English, a short form consent may be used with a COH certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated main consent is processed. However, the research participant is allowed to proceed with surgery/rickham placement and CAR T cell infusion only after the translated main consent form is signed.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies. If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Karnofsky performance status (KPS) >= 60%
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Life expectancy >= 4 weeks
* Participant has a prior histologically-confirmed diagnosis of a grade IV glioblastoma, or has a prior histologically-confirmed diagnosis of a grade II or III malignant brain tumors and now has radiographic progression consistent with a grade IV glioblastoma
* Relapsed disease: radiographic evidence of recurrence/progression of measurable disease after standard therapy, and >= 12 weeks after completion of front-line radiation therapy
* City of Hope (COH) Clinical Pathology confirms matrix metalloproteinase (MMP)2+ tumor expression by immunohistochemistry (>= 20% moderate/high MMP2 [2+/3+])
* No known contraindications to leukapheresis, steroids, or tocilizumab
* White blood cell (WBC) > 2000 /dl (or absolute neutrophil count [ANC] >= 1,000/mm^3) (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Platelets >= 75,000/mm^3 (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Hemoglobin >= 8 g/dl (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Total bilirubin =< 1.5 upper limit of normal (ULN) (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Aspartate aminotransferase (AST) =< 2.5 x ULN (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Alanine aminotransferase (ALT) =< 2.5 x ULN (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Serum creatinine =< 1.6 mg/dL (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Oxygen (O2) saturation >= 95% on room air (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo (to be performed within 14 days prior to leukapheresis unless otherwise stated)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (to be performed within 14 days prior to leukapheresis unless otherwise stated)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of CAR T cells

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior and concomitant therapies
* Owing to higher frequency of wound-related complications, participants who are within 3 months of having received prior bevacizumab therapy at the time of enrollment are excluded.
* Participant has not yet recovered from toxicities of prior therapy
* Other illnesses or conditions
* Uncontrolled seizure activity and/or clinically evident progressive encephalopathy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Active diarrhea
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection
* Other active malignancy
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Noncompliance
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 28 days
  Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 5.0). Rate and associated 90% Clopper and Pearson binomial confidence limits (90% confidence interval) will be estimated for participants experiencing DLTs at the recommended phase 2 dose schedule. Tables will be created to summarize all toxicities and side effects by dose, time post treatment, organ, severity, and arm. 2. Cytokine Release Syndrome (CRS) 3. All other toxicities.

SECONDARY OUTCOMES:
Chimeric antigen receptor (CAR) T cell | 15 years
  Will assess its levels and phenotype detected in tumor cyst fluid (TCF), peripheral blood (PB), and cerebrospinal fluid (CSF) (absolute number per ul by flowcytometry). Statistical and graphical methods will be used.
Endogenous T cell | 15 years
  Will assess its level and phenotype detected in TCF, PB, and CSF (absolute number per ul by flowcytometry). Statistical and graphical methods will be used.
Cytokine levels in TCF, PB and CSF | 15 years
Progression free survival time | At 6 months
Disease response | At 6 months
  Will be assessed by modified Response Assessment in Neuro-Oncology Criteria (RANO) criteria with the need for bevacizumab as an additional indicator of progression.
Overall survival (OS) | At 9 months
  Kaplan Meier methods will be used to estimate median OS and graph the results.
CAR T cells detected in tumor tissue | 15 years
  Will be assessed by immunohistochemistry.
Chlorotoxin-targeted antigen expression levels in tumor tissue | 15 years
  Will assess the pathology H score.
Biomathematical modeling of tumor growth | 15 years
  Will assess perfusion and growth parameters based on serial brain magnetic resonance imaging (MRI)s.

CONTACTS AND LOCATIONS:
Overall Officials: Behnam Badie, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States